CLINICAL TRIAL: NCT03900923
Title: A Phase 2 Study of Cannabidiol as a New Treatment for Autism Spectrum Disorder in Children and Adolescents
Brief Title: Cannabidiol for ASD Open Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-00250
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: ASD; Autism Spectrum Disorder
Keywords: cannabidiol (CBD)
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 98% pure CBD (Experimental): 98% pure CBD. The CBD will be 100mg/mL oral solution provided by Greenwich Biosciences, Inc.
  Interventions: Drug: 98% pure CBD

INTERVENTIONS:
Drug: 98% pure CBD — A Bayesian optimal interval (BOIN) design was used, such that participants were assigned to cohorts of size 3 receiving doses of 3, 6, or 9 mg/kg/day, depending on the treatment response of participants in prior cohorts. The BOIN design has ended, and two doses have been tested and eliminated (3 and 6 mg/kg/day). We are now examining 9 mg/kg/day exclusively.

SUMMARY:
This is a 6-week open trial to identify the optimal dosing of cannabidiol (CBD) in youth with autism spectrum disorder (ASD) and to identify primary and secondary outcomes for future controlled studies. This study evaluates change in symptoms commonly associated with ASD, as evidence suggests that CBD may be eﬀective in addressing diﬃculties such as irritability and anxiety, while maintaining a benign adverse eﬀect (AE) proﬁle in children and adolescents.

30 male and female participants with ASD between the ages of 7 and 17 years old are being recruited. Participants have ﬂuent speech and an estimated IQ greater than or equal to 80. Study intervention is 98% pure CBD. The CBD is Greenwich Biosciences, Inc.'s 100mg/mL oral solution, brand name EPIDIOLEX. First, a Bayesian optimal interval (BOIN) design was used, such that participants were assigned to cohorts of size 3 receiving doses of 3, 6, or 9 mg/kg/day, depending on the treatment response of participants in prior cohorts.

The BOIN design ended after the fifth cohort of participants, and the two lower doses, 3 and 6 mg/kg/day, were eliminated. The highest dose, 9 mg/kg/day, was not tested. Therefore, in subsequent cohorts, we will be examining 9 mg/kg/day exclusively in up to 15 additional participants with co-occurring ASD and attention-deficit/hyperactivity disorder (ADHD) diagnoses, as this clinical profile appears to most closely resemble youth classified as responders within the BOIN design.

ELIGIBILITY:
Inclusion Criteria:

* Male or female pediatric outpatients aged between and including 7 to 17.9 years old
* Diagnosis of ASD confirmed by the ADOS-2 and DSM-5 criteria
* Diagnosis of ADHD confirmed by clinician review of K-SADS-COMP and DSM-5 Criteria
* SRS-2 Total T-score of 66 or higher
* CGI-S score of 4 or higher
* Physical exam and laboratory results that are within normal range for their age
* Fluent speech
* Estimated IQ of at least 80
* Presence of a parent/legal guardian who is able to consent for their participation and complete assessments regarding the child's development and behavior throughout the study

Exclusion Criteria:

* History or current evidence of significantly impaired liver function, defined as 1) Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 5 × upper limit of normal (ULN); 2) ALT or AST > 3 × ULN with concomitant total bilirubin > 2.0 × ULN; or 3) ALT or AST ≥ 3 × ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia
* History of active seizure disorder or epilepsy; patients seizure free for >5 years off of antiepileptic drugs and other than uncomplicated febrile seizures are not excluded
* Exposure to any investigational agent in the 30 days prior to initiation of trial
* Treatment with CBD or other cannabinoid within the previous two months
* Current use of medications metabolized primarily by CYP2B6, CYP2C8, CYP2C9, CYP2C19, CYP3A4, or CYP2D6 isoenzymes. Methylphenidate is not contraindicated.
* History of drug abuse including marijuana/cannabis use in the past 3 months
* Positive urine sample results from drug screening indicating presence of the following drugs: THC, opiates, methamphetamine, or cocaine
* Diagnosis of a known genetic disorder (e.g., Prader-Willi Syndrome, Angelman Syndrome, etc.).
* Active suicidality (ideation and plan) is present
* A current psychiatric diagnosis of bipolar disorder, major depressive disorder (MDD), psychosis, schizophrenia, or post-traumatic stress disorder (PTSD)
* Pregnant or lactating patients or patients who will not agree to be abstinent or use contraception
* A medical condition that severely impacts the subject's ability to participate in the study, interferes with the conduct of the study, confounds interpretation of study results or endangers the subject's well-being
* Diagnosis of Rett Syndrome or Childhood Disintegrative Disorder or marked sensory impairment such as deafness or blindness
* Subjects who have had changes in allied health therapies, behavioral or educational interventions within 4 weeks prior to initiation of trial, other than those associated with school holidays
* Subjects who have had changes in non-exclusionary psychotropic medications within 4 weeks of initiation of trial

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco X Castellanos, MD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in the investigator's University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting requests and accessing data may be found at (Link to be provided).
Access Criteria: Data will be available for any purpose.

RESULTS

PARTICIPANT FLOW:
Groups:
- 3 mg/kg 98% Pure CBD: Participants who received 98% pure CBD: 3 mg/kg/day in Part 1 of the study.
- 6 mg/kg 98% Pure CBD: Participants who received 98% pure CBD: 6 mg/kg/day in Part 1 of the study.
- 9 mg/kg 98% Pure CBD: Participants who received 98% pure CBD: 9 mg/kg/day in Part 2 of the study.
Period: Overall Study
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Started | 6 | 9 | 8
Participants Started Part 1: 3 mg/kg/Day | 6 | 0 | 0
Participants Completed Part 1: 3 mg/kg/Day | 6 | 0 | 0
Participants Started Part 1: 6 mg/kg/Day | 0 | 9 | 0
Participants Completed Part 1: 6 mg/kg/Day | 0 | 9 | 0
Participants Started Part 2: 9 mg/kg/Day | 0 | 0 | 8
Participants Completed Part 2: 9 mg/kg/Day | 0 | 0 | 8
Completed | 6 | 9 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD | Total
Number analyzed (Participants) | 6 | 9 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.32 (2.18) | 11.21 (2.56) | 12.16 (3.4) | 11.31 (2.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 6 | 8 | 8 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4 | 8
  Not Hispanic or Latino | 6 | 4 | 4 | 14
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 3 | 6 | 7 | 16
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression Scale-Improvement (CGI-I)
Description: The physician-rated CGI-I comprises one question asking how much a participant's condition has changed since baseline. The item is answered using a 7-point Likert scale, where 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; and 7 = very much worse. The total score is the item response; lower scores indicate greater improvement.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | 3.17 (0.75) | 2.56 (0.88) | 2.25 (0.71)

2. Secondary Outcome: Change in Repetitive Behavior Scale-Revised (RBS-R) Score
Description: The RBS-R is a 43-item self report used to measure the breadth of repetitive behavior in children. For each item, behaviors are rated on a 4-point scale: 0-Behavior does not occur, 1-Behavior occurs and is a mild problem, 2-Behavior occurs and is a moderate problem, 3-Behavior occurs and is a severe problem. On the last question, participants are asked to "lump together" all of the behaviors described in the questionnaire, and provide a rating for how much of a problem these repetitive behaviors are overall, on a scale from 1-100: 1-Not a problem at all, to 100-As bad as you can imagine. A decrease in scores indicates the repetitive behaviors became less of a problem overall.
  The total score is the sum of all items and ranges from 0 to 229.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | -0.5 (9.52) | -6.67 (9.41) | -4.38 (8.26)

3. Secondary Outcome: Change in Social Responsiveness Scale, 2nd Edition (SRS-2), School-Age Form Score
Description: The SRS-2 is a 65-item questionnaire assessing Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted Interests and Repetitive Behavior. Items are scored on a 4-point scale (ranging from 1=not true to 4=almost always true). The raw score is the sum of responses and is converted to a T-score; the final T-score has a mean of 50 points with a standard deviation of 10 points, where lower scores indicate greater social responsiveness:
  * Less than or equal to 59 = Low-to-no symptom impacts
  * Between 60-65 = Mild-to-moderate defcits in social interaction
  * Between 66-75 = Moderate defcit in social interaction
  * Greater than or equal to 76 = Severe
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | -6.17 (5) | -14 (12.55) | -17.4 (5.5)

4. Secondary Outcome: Change in Aberrant Behavior Checklist (ABC) - Irritability Subscale Score
Description: The ABC Irritability subscale comprises 15 items rated on a 4-point scale (ranging from 0=no problem at all to 3 = problem is severe in degree). The total score is the sum of responses and ranges from 0 to 45; higher scores indicate greater presences of irritability related behavior.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | -5.5 (5.4) | -5.89 (7.51) | -1.4 (3.1)

5. Secondary Outcome: Change in Screen for Child Anxiety Related Disorders (SCARED), Parent Version Score
Description: The SCARED, Parent Version is a 41-item parent-report measure developed to measure child anxiety symptoms. Subscales include Somatic Symptoms/Panic Disorder, Generalized Anxiety Disorder, Separation Anxiety, Social Phobia, and School Phobia. Items are rated on a 3-point scale ranging from 0=not true or hardly ever true to 2=very true or often true. The total score is the sum of responses and ranges from 0 to 82; lower scores indicate lesser child anxiety symptoms.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | -6.33 (13.7) | -16 (17.12) | -3.25 (12.6)

6. Secondary Outcome: Change in Sleep Disturbance Scale for Children (SDSC) Score
Description: The SDSC is a 26-item parent-completed assessment of their child's sleep-wake rhythm. The questionnaire measures Disorders of Initiating and Maintaining Sleep, Sleep Breathing Disorders, Disorders of Arousal, Sleep Wake Transition Disorders, Disorders of Excessive Somnolence, and Sleep Hyperhydrosis. Items are rated on 5-point scale where 1=never and 5=always (daily). The total score is the sum of responses and ranges from 26 to 130; lower scores indicate healthier sleep-wake rhythms.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | -7.5 (12.65) | -6.89 (5.44) | -0.13 (4.82)

7. Secondary Outcome: Change in Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) Parent/Caregiver Form Score
Description: Used to measure adaptive functioning across three core domains (Communication, Daily Living Skills, and Socialization), and two optional domains (Motor Skills and Maladaptive Behavior); items are rated on a 3-point scale (0=never; 1=sometimes; 2=usually or often). The core domains sum to a total Adaptive Behavior Composite. The range of possible composite scores ranges from 20-140, with a higher score indicating higher levels of adaptive functioning.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | -0.5 (3.89) | 4.33 (5.72) | 8.88 (7.32)

8. Secondary Outcome: Change in Clinical Global Impression-Severity (CGI-S) Score
Description: 1-item assessment of clinicians impression of severity of illness. Illness severity is rated on a 7-point scale ranging from 1=not at all to 7=among the most extremely ill.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | -0.5 (0.84) | -1 (0.87) | -0.5 (0.53)

9. Secondary Outcome: Change in Autism Family Experience Questionnaire (AFEQ) Score
Description: Parent/Caregiver form used to measure impact of autism interventions on family experience and quality of life. Items are rated on a 5-point scale where 1=always and 5=never. The total score is the sum of responses and ranges from 48 - 240; lower scores indicate better outcomes.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | -3.17 (14.5) | -14 (20.1) | -8.88 (8.37)

10. Secondary Outcome: Change in Anxiety Scale for Children - Autism Spectrum Disorder - Parent Versions (ASC-ASD-P) Score
Description: 24-item Parent/Caregiver-completed form developed to detect symptoms of anxiety in youth with ASD. Items are rated on a 4-point scale (0=never and 3=always). The total score is the sum of responses and ranges from 0 to 72; lower scores indicate lesser symptoms of anxiety.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | -2.33 (4.76) | -6.56 (9.84) | -3.13 (6.15)

11. Secondary Outcome: Anxiety Scale for Children - Autism Spectrum Disorder (ASC-ASD-C) - Child Version
Description: 24-item Child-completed form developed to detect symptoms of anxiety in youth with ASD. Items are rated on a 4-point scale (0=never and 3=always). The total score is the sum of responses and ranges from 0 to 72; lower scores indicate lesser symptoms of anxiety.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | -4 (6.81) | -4.78 (5.61) | -6.5 (11.2)

12. Secondary Outcome: Change in Ohio State University (OSU) Autism Clinical Global Impressions: Severity
Description: Reflects clinicians impression of severity of illness on a 7-point scale ranging from 1=not present to 7="classic" autism.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | 0 (0) | -0.22 (0.67) | -0.38 (0.52)

13. Secondary Outcome: OSU Autism Clinical Global Impressions: Improvement
Description: Reflects clinicians impression of improvement on a 7-point scale ranging from 1=very much improved to 7=very much worse.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | 3.67 (0.82) | 2.78 (0.67) | 2.38 (0.52)

14. Secondary Outcome: Change in Behavioral Inflexibility Scale (BIS) Score
Description: 38-item Parent/Caregiver-completed measure designed to assess rigid patterns of behavior commonly associated with ASD. Items are rated on a 6-point Likert scale where 0=Not at all a problem and 5=Very severe or extreme problem. The total score is the sum of responses and ranges from 0 to 228; higher scores indicate greater behavioral inflexibility.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | -13 (28.61) | -25.4 (40.54) | -9.75 (13.73)

15. Secondary Outcome: Change in Home Situations Questionnaire - Modified for ASD (HSQ-ASD) Score
Description: 24-item Parent/Caregiver-completed questionnaire measuring behavioral noncompliance in everyday settings over the past four weeks. Severity of non-compliance is rated on a 9-point Likert scale (where 1 = no interruption, and 9 = frequent/consistent interruption). The total score is the sum of responses and ranges from 24 to 216; higher scores indicate greater behavioral noncompliance.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 6 | 9 | 8
score on a scale | -8.67 (40.51) | -23.67 (20.02) | -5.88 (6.73)

16. Secondary Outcome: Change in Strengths and Weaknesses of Attention-Deficit/Hyperactivity Disorder Symptoms and Normal Behavior (SWAN) Score
Description: SWAN is an 18-item Parent/Caregiver-completed measure designed to assess symptoms of ADHD in children and adolescents. Items are rated on a 7-point Likert scale, where Far Below Average = 3, Below Average = 2, Somewhat Below Average = 1, Average = 0, Somewhat Above Average = -1, Above Average = -2, and Far Above Average = -3. The total score is the sum of responses and ranges from -54 to 54; the lower the score, the higher the severity of ADHD symptoms.
Time Frame: Baseline, Week 6
Population: This outcome was not analyzed/assessed among participants in Part 1 of the trial (3 mg/kg and 6 mg/kg CBD arms).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
Number analyzed (Participants) | 0 | 0 | 7
score on a scale |  |  | -2.71 (8.08)

ADVERSE EVENTS:
Time Frame: 6 weeks after participant received first dose.
Description: PI monitor for adverse events (AEs) at each follow-up visit. Study coordinator phone call to parents/caregivers to assess for AEs at weeks 1, 3, and 5. Participants and caregivers completed UKU Side Effects Rating Scale at weeks 2, 4, and 6. Participants were not assessed for all-cause mortality.
Arm/Group | 3 mg/kg 98% Pure CBD | 6 mg/kg 98% Pure CBD | 9 mg/kg 98% Pure CBD
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 6/6 | 8/9 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3 mg/kg 98% Pure CBD (N=6) | 6 mg/kg 98% Pure CBD (N=9) | 9 mg/kg 98% Pure CBD (N=8)
Palpitations/Tachycardia (Cardiac disorders) | 0 | 0 | 2
Increased Salivation (Endocrine disorders) | 1 | 2 | 4
Dry mouth (Endocrine disorders) | 1 | 0 | 1
Increased sweating (Endocrine disorders) | 1 | 0 | 1
Appetite increase (Gastrointestinal disorders) | 0 | 0 | 2
Appetite decrease (Gastrointestinal disorders) | 0 | 2 | 1
Weight gain (General disorders) | 1 | 0 | 1
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Akathesia (Nervous system disorders) | 1 | 2 | 3
Dystonia (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 0
Increased stereotypies (Nervous system disorders) | 0 | 2 | 0
Paresthesias (Nervous system disorders) | 1 | 1 | 1
Rigidity (Nervous system disorders) | 1 | 1 | 0
Asthenia (Psychiatric disorders) | 2 | 2 | 0
Apathy (Psychiatric disorders) | 0 | 2 | 0
Concentration difficulties (Psychiatric disorders) | 0 | 1 | 2
Depressed Mood (Psychiatric disorders) | 1 | 1 | 0
Emotionality (Psychiatric disorders) | 0 | 3 | 0
Oppositionality (Psychiatric disorders) | 2 | 0 | 0
Increased sleep duration (Psychiatric disorders) | 1 | 4 | 4
Decreased sleep duration (Psychiatric disorders) | 1 | 2 | 1
Sleepiness/Sedation (Psychiatric disorders) | 3 | 2 | 1
Heavier Sleep (Psychiatric disorders) | 1 | 1 | 1
Increased Dream Activity (Psychiatric disorders) | 1 | 3 | 4
Sleep-onset Insomnia (Psychiatric disorders) | 0 | 2 | 1
Polyuria (Renal and urinary disorders) | 1 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT03900923/Prot_SAP_000.pdf